CLINICAL TRIAL: NCT06330220
Title: Optical Coherence Tomography Angiography and Microperimetry After Aflibercept in Wet Age-related Macular Degeneration Patients With the Better Baseline Visual Acuity (≥20/40)
Brief Title: Visual Function Change in Wet Age-related Macular Degeneration Patients With Better Baseline Visual Acuity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chang Ki Yoon, Clinical Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-015-1161
Record Dates: First submitted 2024-03-07; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aflibercept loading (Experimental): Administration of 2㎎ intravitreal aflibercept three times monthly after diagnosis
  Interventions: Drug: Aflibercept Injection [Eylea]

INTERVENTIONS:
Drug: Aflibercept Injection [Eylea] — intravitreal injection
  Other Names: Eylea injection

SUMMARY:
Although the number of wet AMD patients with the better visual acuity is increasing, the visual improvement in patients with the better vision may not be so significant after anti-vascular endothelial growth factor (VEGF) treatments because of 'ceiling effect'. The aim of current study is to investigate the improvement of visual function after aflibercept treatments using microperimetry in wet AMD patients with the better baseline visual acuity (≥20/40).

DETAILED DESCRIPTION:
This study is designed to show the clinical effect of aflibercept in early disease course for wet age-related macular degeneration (AMD) with better visual acuity. It is important to extend the usage of aflibercept and give the treatment chance to patient.

VIEW 1 and VIEW 2 Study demonstrated that aflibercept was excellent treatment for choroidal neovascularization secondary to AMD, but the study enrolled patients with a range of visual acuity (20/40 to 20/320). A previous study with ranibizumab, Marina and Anchor studies also had the same inclusion criteria with VIEW studies. Recently, the number of wet AMD patients with the better visual acuity is increasing. However, the visual improvement in patients with the better vision may not be so significant after anti-vascular endothelial growth factor (VEGF) treatments because of 'ceiling effect'.

The aim of current study is to investigate the improvement of visual function after aflibercept treatments using microperimetry in wet AMD patients with the better baseline visual acuity (≥20/40). And correlation of optical coherence tomography angiography (OCTA) findings and microperimetry will be evaluated to provide investigators with additional data about the effects of therapeutic agents.

In this study, the aflibercept will be treated according to the Ministry of Food and drug safety guideline. Also, the patients will be provided with aflibercept, microperimetry and imaging tests (fluorescein angiography, indocyanine green angiography, optical coherence tomography and OCTA).

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or older than 50 years
* Treatment Naïve with active subfoveal choroidal neovascularization (CNV) lesion secondary to age-related macular degeneration (AMD) in the study eye
* Baseline visual acuity equal to or better than 20/40
* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Willingness and ability to undertake all scheduled visits and assessments

Exclusion Criteria:

* Sub- or intra-retinal hemorrhage that comprises more than 50% of the entire lesion in the study eye
* Scar, fibrosis or atrophy involving the center of the fovea in the study eye
* Presence of CNV in either eye due to other causes, such as ocular histoplasmosis, trauma, multifocal choroiditis, angioid streaks, history of choroidal rupture or pathologic myopia
* Presence of retinal pigment epithelial tears or rips involving the macula in the study eye
* Presence of macular hole at any stage in the study eye
* Any concurrent macular abnormality other than AMD in the study eye including epiretinal membrane, macular telangiectasia, retinal vascular abnormality.
* History of intraocular surgery except cataract operation
* Any previous intravitreal treatment to treat neovascular AMD in study eye.
* Spherical equivalent of the refractive error in the study eye demonstrating more than 8 diopters of myopia
* Presence of glaucoma that affect visual field in the study eye
* Uncontrolled ocular hypertension in the study eye (defined as intraocular pressure ≥ 25 mg despite treatment with anti-glaucoma medication) in the study eye
* History of allergy to the fluorescein sodium for injection in angiography
* History or clinical evidence of diabetic retinopathy much severe than mild non-proliferative diabetic retinopathy or diabetic macular edema in either eye
* Stroke, transient ischemic attacks, or myocardial infarction within 90 days prior to screening
* Prior treatment involving macula with photodynamic therapy with verteporfin, transpupillary thermotherapy, radiation therapy, or retinal laser treatment in the study eye, and such medications will not be allowed during the study period.
* Current use of systemic medications known to be toxic to the lens, retina or optic nerve, including deferoxamine, chloroquine/hydroxychloroquine, tamoxifen, phenothiazines, vigabatrin and ethambutol, and such medications will not be allowed during the study period.
* Patients incapable of performing diagnostic tests for reasons including physical or attention limitation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Retinal sensitivity change after aflibercept treatment using microperimetry in wet age-related macular degeneration patients | 12 weeks
  Visual function changes by assessing retinal sensitivity changes using microperimetry after aflibercept loading injection in wet age-related macular degeneration patients

SECONDARY OUTCOMES:
The correlation of OCT and OCT angiography parameters with retinal sensitivity change measured by microperimetry | 12 weeks
  OCT and OCT angiography parameters associated with retinal sensitivity change

CONTACTS AND LOCATIONS:
Overall Officials: Chang Ki Yoon, Ph.D, Principal Investigator — Seoul National University College of Medicine, Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea